CLINICAL TRIAL: NCT05957705
Title: Maxillary Sinus Augmentation With Xenogeneic Bone Graft Associated or Not With Fibrin Rich in Platelets and Leukocytes Produced by Horizontal Centrifugation for Early Implant Placement: a Randomized Controlled Split-mouth Clinical Trial.
Brief Title: Maxillary Sinus Augmentation With Xenogeneic Bone Graft Associated or Not With Fibrin Rich in Platelets and Leukocytes Produced by Horizontal Centrifugation: A Randomized Clinical Trial.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Michel Reis Messora, Associate professor at the department of Oral and Maxillofacial Surgery and Periodontology, School of Dentistry of Ribeirao Preto, University of Sao Paulo-USP, Ribeirao Preto, São Paulo, Brazil, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 29428820.3.0000.5419
Record Dates: First submitted 2023-07-15; First posted 2023-07-24 (Actual); Last update posted 2023-07-24 (Actual); Status verified 2023-07

CONDITIONS: Platelet-rich Fibrin; Sinus Floor Augmentation; Cone-beam Computed Tomography; Dental Implants; Bone Substitutes; Maxillary Sinus; Atrophic Maxilla
MeSH Terms: conditions — Atrophic Maxilla | interventions — Dental Implants

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: The researchers responsible for the tomographic and histometric analysis will not be aware of the type of group in which the sample is located.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Bilateral Sinus Augmentation (Active Comparator): Split-mouth bilateral sinus augmentation of xenogeneic bone graft associated or not with platelet-rich fibrin produced by horizontal centrifugation.
  Interventions: Procedure: Maxilar Sinus augmentation
- Early dental implant placement by Guided Surgery (Active Comparator)
  Interventions: Procedure: Dental implant placement using guided surgery
- Dental implants reopening surgery for implant load (Active Comparator)
  Interventions: Procedure: Dental implant placement using guided surgery

INTERVENTIONS:
Procedure: Maxilar Sinus augmentation — The patients will be submitted to bilateral sinus augmentation using two different techniques to provide enough bone tissue for dental implants placement.
  Other Names: Maxilar sinus lift; Maxilary sinus lifting
  Arms: Bilateral Sinus Augmentation
Procedure: Dental implant placement using guided surgery — After 4 months of sinus augmentation, patients will be prepared to receive dental implants for oral rehabilitation. Performed by guided surgery the implants will be placed at the best location for the rehabilitation and at the place were the sinus lighting were performed.
  Other Names: Dental implant; Dental implant surgery; Dental implant guided surgery
  Arms: Dental implants reopening surgery for implant load; Early dental implant placement by Guided Surgery

SUMMARY:
The objective of study is to evaluate the influence of the use of Platelet Rich Fibrin (PRF) from the patient's produced by a new horizontal centrifugation protocol associated with particulate xenogenous bone graft in the rehabilitation of atrophic maxillary sinus for early osseointegrated implants plancement. In a split-mouth model, twelve patients in need of rehabilitation with at least two bilateral implants in the regions of atrophic maxillary sinus will simultaneously undergo bone reconstruction using deproteinized particulate xenogenous bone (Bio-Oss Small®; Geistlich AG, Wolhusen , Switzerland). Randomly, one of the surgical sites of each patient will be reconstructed using the associated technique of solid PRF + Liquid PRF with the xenogen material, where at the end of the grafting procedure, both sites will be protected by a collagen membrane (Bio-Gide® Compressed; Geistlich AG, Wolhusen, Switzerland) positioned over the surgical access of the maxillary sinus. During the research, cone-beam computed tomography scans will be performed preoperatively, immediately after surgical procedure, 3 months after maxillary sinus reconstruction, after immediate implants placement and 12 months after functional load of the implants for comparative volume measurement of tissue gain and the maintenance of the grafted tissue. During the implant surgery, bilateral biopsies will be collected after 4 months of the regenerative surgical procedure during the early dental implants surgery by virtually guided surgery. The stability of the implants will be measured by means of resonance frequency analysis (ISQ) after the immediate postoperative period and 6 postoperative months as the clinical success rates of the implants after 12 months with functional load. The tissue samples will be used for histological, histomorphometric, immunohistochemistry and microtomographic analysis. All data obtained will be statistically analyzed.

ELIGIBILITY:
Inclusion Criteria:

* need of at least one dental implant in atrophic maxillary sinus region;
* insufficient amount of vertical bone remnant for the dental implants surgery (maximum of 4mm);
* sufficient horizontal bone thickness for dental implants rehabilitation;
* present edentulism in the area to be treated for at least 6 months;
* similar pattern of pneumatization of the maxillary sinuses.

Exclusion Criteria:

* any contraindication for the installation of dental implants;
* need of horizontal bone augmentation;
* pacientes with inflammatory or autoimmune disease in the oral cavity;
* use of immunosuppressants, corticosteroids or bisphosphonates for medical needs;
* pacientes with history of malignancy in the last 5 years;
* smoking patients or patients reporting excessive alcohol consumption;
* decompensated systemic condition, uncontrolled periodontal disease, insulin-dependent diabetic patients, patients with blood-related diseases and patients who need oral rehabilitation in the lower arch;
* It is also noteworthy that patients with a history of reconstructive bone therapies in the maxillary sinus region or with a history of oroantral communication will be excluded from this research.

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2021-03-17 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
Micro-CT and Histometric analyses | 4 Months
  After the period of 4 months from sinus reconstructions, during the dental implant placement by guided surgery, bone samples will be collected at the same location of the implants preparation. The collected bone tissue will be prepared and submitted to Micro-CT and histometric analyses.

SECONDARY OUTCOMES:
Dental Implants ISQ measurement | 6 months
  ISQ will be measured at the moment of implant placement and after 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Michel R Messora, Phd, Study Chair — Universidade de São Paulo - FORP-USP; Gabriel GD Reis, Phd Student, Principal Investigator — Universidade de São Paulo - FOR-USP
Locations (1):
- School of Dentistry of Ribeirão Preto - USP, Ribeirão Preto, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Undecided